CLINICAL TRIAL: NCT01194973
Title: An Open-label, Multi-center Clinical Trial of Eculizumab in Adult Patients With Atypical Hemolytic-uremic Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C10-004
Record Dates: First submitted 2010-08-31; First posted 2010-09-03 (Estimated); Results first posted 2015-04-24 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2015-04

CONDITIONS: Atypical Hemolytic-Uremic Syndrome
Keywords: Atypical Hemolytic-Uremic Syndrome
MeSH Terms: conditions — Atypical Hemolytic Uremic Syndrome | interventions — eculizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Eculizumab (Experimental)
  Interventions: Drug: Eculizumab

INTERVENTIONS:
Drug: Eculizumab — All patients received open-label eculizumab administered intravenously on the following dose schedule: Induction dose - 900 mg per week for four weeks and a dose of 1200 mg one week later; Maintenance dose - 1200 mg every two weeks. Patients who received plasma exchange or infusion during the eculizumab treatment period received a supplemental dose of 600 mg within one hour before plasma infusion or within one hour after the completion of each plasma exchange.

SUMMARY:
The record Primary purpose is to assess the efficacy of eculizumab in adult patients with Atypical Hemolytic- Uremic Syndrome (aHUS) to control Thrombotic Microangiopathy (TMA) as characterized by thrombocytopenia, hemolysis and renal impairment.

ELIGIBILITY:
Inclusion:

1. Patient must be willing and able to give written informed consent.
2. Patient's age > 18 years.
3. Patients exhibit thrombocytopenia, hemolysis and elevated Serum Creatinine.
4. Patients with diagnosis of aHUS with or without an identified complement regulatory protein genetic abnormality or anti-complement factor antibody and for whom etiologies of hemolytic uremic syndrome have been ruled out as confirmed in the exclusion criteria
5. Female patients of childbearing potential must be practicing an effective, reliable and medically approved contraceptive regimen during the entire duration of the study, including the follow-up period. At the time of the last follow-up visit, patients must agree to continue to use adequate contraception methods for up to 5 months following discontinuation of eculizumab treatment.
6. Able and willing to comply with study procedures

Exclusion:

1. Chronic dialysis.
2. Prior eculizumab use or hypersensitivity to eculizumab, to murine proteins or to one of the excipients.
3. Known familial a disintegrin and metalloproteinase with a thrombospondin type 1 motif, member 13 (ADAMTS-13) deficiency (ADAMTS-13 <5%).
4. Typical Hemolytic-Uremic Syndrome (HUS) (known Shiga toxin +).
5. History of malignancy within 5 years of screening.
6. Known human immunodeficiency virus (HIV) infection.
7. Identified drug exposure-related hemolytic-uremic syndrome (HUS).
8. Infection-related HUS.
9. HUS related to bone marrow transplant (BMT).
10. HUS related to vitamin B12 deficiency.
11. Known Systemic Lupus Erythematosus (SLE) or antiphospholipid antibody positivity or syndrome.
12. Patients with a confirmed diagnosis of sepsis defined as positive blood cultures within 7 days of the screening visit and not treated with antibiotics to which the organism is sensitive.
13. Presence or suspicion of active and untreated systemic bacterial infection that, in the opinion of the Investigator confounds an accurate diagnosis of aHUS or impedes the ability to manage the aHUS disease.
14. Pregnancy or lactation.
15. Unresolved systemic meningococcal disease.
16. Any medical or psychological condition that, in the opinion of the investigator, could increase the patient's risk by participating in the study or confound the outcome of the study.
17. Patients receiving chronic intravenous immunoglobulin (IVIg) within 8 weeks or chronic Rituximab therapy within 12 weeks of screening visit.
18. Patients receiving other immunosuppressive therapies such as steroids, mechanist target of rapamycin (mTOR) inhibitors, calcineurin inhibitors (e.g., cyclosporine or tacrolimus) are excluded unless: [1] part of an established post-transplant anti-rejection regime, or [2] patient has confirmed anti-Complement Factor Antibodies requiring immunosuppressive therapy, or [3] steroids are being used for a condition other than aHUS (example asthma).
19. Participation in any other investigational drug trial or device trial, or procedures beginning 4 weeks prior to screening and throughout the entire trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2010-07; Primary Completion 2013-10 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (22):
- United States (5):
  - Burlington, Massachusetts
  - Hackensack, New Jersey
  - New York, New York
  - Columbus, Ohio
  - Houston, Texas
- Liège, Belgium
- France (7):
  - Caen
  - Lille
  - Nantes
  - Nice
  - Paris
  - Toulouse
  - Tours
- Germany (2):
  - Essen
  - Hanover
- Italy (2):
  - Bergamo
  - Florence
- Spain (2):
  - Barcelona
  - Córdoba
- United Kingdom (3):
  - Exeter
  - London
  - Newcastle

REFERENCES:
- [Derived] Pugh D, O'Sullivan ED, Duthie FA, Masson P, Kavanagh D. Interventions for atypical haemolytic uraemic syndrome. Cochrane Database Syst Rev. 2021 Mar 23;3(3):CD012862. doi: 10.1002/14651858.CD012862.pub2. PMID 33783815
- [Derived] Cofiell R, Kukreja A, Bedard K, Yan Y, Mickle AP, Ogawa M, Bedrosian CL, Faas SJ. Eculizumab reduces complement activation, inflammation, endothelial damage, thrombosis, and renal injury markers in aHUS. Blood. 2015 May 21;125(21):3253-62. doi: 10.1182/blood-2014-09-600411. Epub 2015 Apr 1. PMID 25833956

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 44 patients diagnosed with aHUS signed the informed consent and of these, 41 patients were treated. Three patients were excluded from the study due to failed screening procedure and did not receive eculizumab.
Pre-assignment Details: At screening, patients had to have signs or symptoms of hemolysis; serum creatinine level ≥ ULN and platelet count < LLN
Period: Screening Period
Arm/Group | Eculizumab
Started | 44
Completed | 41
Not Completed | 3
Not completed — Screen Failure | 3
Period: 26 Week Treatment Period
Arm/Group | Eculizumab
Started | 41
Completed | 38
Not Completed | 3
Not completed — Adverse Event | 1
Not completed — Lack of Efficacy | 1
Not completed — Pregnancy | 1

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) population was defined as all patients who received any amount of eculizumab, and were considered evaluable for safety and efficacy analyses. For both the efficacy and safety analyses, all 41 patients who were treated with study drug were included in the ITT population.
Arm/Group | Eculizumab
Number analyzed (Participants) | 41
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.3 (15.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 38
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Complete TMA Response
Description: Proportion of Patients with Complete TMA response was determined and defined by normalization of hematological parameters (platelet count and LDH) and preservation of renal function (defined as < 25% increase in serum creatinine from baseline) which were sustained for at least two consecutive measurements obtained at least four weeks apart.
Time Frame: Through 26 weeks
Population: The tabulations of the proportions of patients with Complete TMA Response through 26 weeks were performed for the ITT population. Exact binomial two-sided 95% CI using the Clopper-Pearson method for the responder rate was presented.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Eculizumab
Number analyzed (Participants) | 41
Percentage of Participants | 73.2 [57.1 to 85.8]

2. Primary Outcome: Percentage of Patients With Modified Complete TMA Response
Description: Proportion of Patients with Modified Complete TMA response through 26 weeks of treatment was determined and defined by normalization of hematological parameters (platelet count and LDH) and improvement in renal function (defined as ≥ 25% reduction from the baseline value in serum creatinine, which were sustained for at least two consecutive measurements obtained at least four weeks apart.
Time Frame: Through 26 weeks
Population: The tabulations of the proportions of patients with Modified Complete TMA Response through 26 weeks were performed for the ITT population. Exact binomial two-sided 95% CI using the Clopper-Pearson method for the responder rate was presented.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Eculizumab
Number analyzed (Participants) | 41
Percentage of Participants | 56.1 [39.7 to 71.5]

3. Secondary Outcome: Percentage of Patients With Complete Hematologic Response
Description: Proportion of Patients with Complete Hematologic response through end of study was determined and defined by normalization of platelet count and LDH sustained for at least two consecutive measurements obtained at least four weeks apart.
Time Frame: Through 26 weeks
Population: The tabulations of the proportions of patients with Complete Hematologic Response through 26 weeks were performed for the ITT population. The number of patients with response and responder rate, along with an exact two-sided 95% CI were summarized.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Eculizumab
Number analyzed (Participants) | 41
Percentage of Participants | 87.8 [73.8 to 95.9]

4. Secondary Outcome: Percentage of Patients With Platelet Count Normalization
Description: Proportion of Patients with Platelet Count Normalization through 26 weeks of treatment was determined and defined as the platelet count observed to be ≥ 150 x 109/L on at least two consecutive measurements which span a period of at least four weeks
Time Frame: Through 26 weeks
Population: The tabulations of the proportions of patients with Platelet Count Normalization through 26 weeks were performed for the ITT population. The number of patients with response and responder rate, along with an exact two-sided 95% CI were summarized.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Eculizumab
Number analyzed (Participants) | 41
Percentage of Participants | 97.6 [87.1 to 99.9]

5. Secondary Outcome: Percentage of Patients With Estimated Glomerular Filtration Rate (eGFR) Improvement
Description: Proportion of Patients with Estimated Glomerular Filtration Rate (eGFR) Improvement was determined and defined as an increase in eGFR by ≥ 15 mL/min/1.73m^2 from baseline, sustained for at least two consecutive measurements obtained at least four weeks apart.
Time Frame: Through 26 weeks
Population: The tabulations of the proportions of patients with Estimated Glomerular Filtration Rate (eGFR) Improvement through 26 weeks were performed for the ITT population. The number of patients with response and responder rate, along with an exact two-sided 95% CI were summarized.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Eculizumab
Number analyzed (Participants) | 41
Percentage of Participants | 53.7 [37.4 to 69.3]

6. Secondary Outcome: Platelet Count Change From Baseline to 26 Weeks
Time Frame: Through 26 weeks
Population: Change from baseline platelet counts were analyzed for the ITT population using a repeated measures Analysis of variance (ANOVA) model. The estimated LS means of change from baseline at each post-baseline visit alongside with 95% CIs and P-values were calculated, as were the parameter estimates for the covariates and their associated P-values.
Measure: Least Squares Mean (95% Confidence Interval); unit: 10^9 cells/L
Arm/Group | Eculizumab
Number analyzed (Participants) | 41
10^9 cells/L | 117.68 [92.77 to 142.59]
Statistical Analysis 1: Comparison: Eculizumab; Test type: Superiority or Other; p < 0.0001, ANOVA; LS mean change from baseline = 117.68, 95% CI 2-sided [92.77 to 142.59]

7. Secondary Outcome: Percentage of Patients With Complete TMA Response
Description: Proportion of Patients with Complete TMA response through end of study was determined and defined by normalization of hematological parameters (platelet count and LDH) and preservation of renal function (defined as < 25% increase in serum creatinine from baseline) which were sustained for at least two consecutive measurements obtained at least four weeks apart.
Time Frame: Through End of Study, Median Exposure 52 Weeks
Population: The tabulations of the proportions of patients with Complete TMA Response through end of study were performed for the ITT population. Exact binomial two-sided 95% CI using the Clopper-Pearson method for the responder rate was presented.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Eculizumab
Number analyzed (Participants) | 41
Percentage of Participants | 80.5 [65.1 to 91.2]

8. Secondary Outcome: Percentage of Patients With Modified Complete TMA Response
Description: Proportion of Patients with Modified Complete TMA response through end of study was determined and defined by normalization of hematological parameters (platelet count and LDH) and improvement in renal function (defined as ≥ 25% reduction from the baseline value in serum creatinine, which were sustained for at least two consecutive measurements obtained at least four weeks apart.
Time Frame: Through End of Study, Median Exposure 52 Weeks
Population: The tabulations of the proportions of patients with Modified Complete TMA Response through end of study were performed for the ITT population. Exact binomial two-sided 95% CI using the Clopper-Pearson method for the responder rate was presented.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Eculizumab
Number analyzed (Participants) | 41
Percentage of Participants | 63.4 [46.9 to 77.9]

9. Secondary Outcome: Percentage of Patients With Complete Hematologic Response
Description: Proportion of Patients with Complete Hematologic response through end of study of treatment was determined and defined by normalization of platelet count and LDH sustained for at least two consecutive measurements obtained at least four weeks apart.
Time Frame: Through End of Study, Median Exposure 52 Weeks
Population: The tabulations of the proportions of patients with Complete Hematologic Response through end of study were performed for the ITT population. The number of patients with response and responder rate, along with an exact two-sided 95% CI were summarized.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Eculizumab
Number analyzed (Participants) | 41
Percentage of Participants | 97.6 [87.1 to 99.9]

10. Secondary Outcome: Percentage of Patients With Platelet Count Normalization
Description: Proportion of Patients with Platelet Count Normalization through end of study of treatment was determined and defined as the platelet count observed to be ≥ 150 x 109/L on at least two consecutive measurements which span a period of at least four weeks
Time Frame: Through End of Study, Median Exposure 52 Weeks
Population: The tabulations of the proportions of patients with Platelet Count Normalization through end of study were performed for the ITT population. The number of patients with response and responder rate, along with an exact two-sided 95% CI were summarized.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Eculizumab
Number analyzed (Participants) | 41
Percentage of Participants | 100.0 [91.4 to 100.0]

11. Secondary Outcome: Percentage of Patients With Estimated Glomerular Filtration Rate (eGFR) Improvement
Description: Proportion of Patients with Estimated Glomerular Filtration Rate (eGFR) Improvement was determined and defined as an increase in eGFR by ≥ 15 mL/min/1.73m^2 from baseline sustained for at least two consecutive measurements obtained at least four weeks apart
Time Frame: Through End of Study, Median Exposure 52 Weeks
Population: The tabulations of the proportions of patients with Estimated Glomerular Filtration Rate (eGFR) Improvement through end of study were performed for the ITT population. The number of patients with response and responder rate, along with an exact two-sided 95% CI were summarized for each parameter.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Eculizumab
Number analyzed (Participants) | 41
Percentage of Participants | 61.0 [44.5 to 75.8]

12. Secondary Outcome: Platelet Count Change From Baseline to 52 Weeks
Time Frame: Through 52 Weeks
Population: Change from baseline platelet counts were analyzed for the ITT population using a repeated measures ANOVA model. The estimated LS means of change from baseline at each post-baseline visit alongside with 95% CIs and P-values were calculated, as were the parameter estimates for the covariates and their associated P-values.
Measure: Least Squares Mean (95% Confidence Interval); unit: 10^9 cells/L
Arm/Group | Eculizumab
Number analyzed (Participants) | 41
10^9 cells/L | 102.49 [68.15 to 136.82]
Statistical Analysis 1: Comparison: Eculizumab; Test type: Superiority or Other; p < 0.0001, ANOVA; LS mean change from baseline = 102.49, 95% CI 2-sided [68.15 to 136.82]

ADVERSE EVENTS:
Time Frame: Through end of study; exposure to eculizumab in this study extended for a median duration of 11.9 months and ranged from 2.9 months to 28.8 months
Description: At every visit, patients were asked a standard non-leading question to elicit any changes in their medical well-being including inquiry about any hospitalization, accidents and new or changed concomitant medication regimens. AEs were also documented from any data collected (e.g. laboratory values, physical examination findings, ECG changes, etc.)
Arm/Group | Eculizumab
Serious Adverse Events (participants affected / at risk) | 19/41
Other Adverse Events (participants affected / at risk) | 41/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eculizumab (N=41)
Haemolytic uraemic syndrome (Blood and lymphatic system disorders) | 1
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Medical device complication (General disorders) | 1
Kidney transplant rejection (Immune system disorders) | 1
Bronchitis (Infections and infestations) | 1
Device related infection (Infections and infestations) | 1
Device related sepsis (Infections and infestations) | 2
Genitourinary tract gonococcal infection (Infections and infestations) | 1
Meningitis meningococcal (Infections and infestations) | 1
Meningococcal sepsis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 2
Shunt infection (Infections and infestations) | 1
Shunt malfunction (Injury, poisoning and procedural complications) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Convulsion (Nervous system disorders) | 2
Haemorrhage intracranial (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 1
Renal failure acute (Renal and urinary disorders) | 2
Renal failure chronic (Renal and urinary disorders) | 2
Renal impairment (Renal and urinary disorders) | 2
Renal vessel disorder (Renal and urinary disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Rash papular (Skin and subcutaneous tissue disorders) | 1
Skin necrosis (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 1
Hypertensive crisis (Vascular disorders) | 1
Venous thrombosis (Vascular disorders) | 1
Hypoglycemia (Metabolism and nutrition disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eculizumab (N=41)
ANAEMIA (Blood and lymphatic system disorders) | 7
EOSINOPHILIA (Blood and lymphatic system disorders) | 1
IRON DEFICIENCY ANAEMIA (Blood and lymphatic system disorders) | 1
LEUKOPENIA (Blood and lymphatic system disorders) | 5
LYMPHOPENIA (Blood and lymphatic system disorders) | 3
NEUTROPENIA (Blood and lymphatic system disorders) | 2
SPONTANEOUS HAEMATOMA (Blood and lymphatic system disorders) | 1
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 2
ANGINA PECTORIS (Cardiac disorders) | 1
CARDIOMYOPATHY (Cardiac disorders) | 1
PALPITATIONS (Cardiac disorders) | 1
TACHYCARDIA (Cardiac disorders) | 2
EAR PAIN (Ear and labyrinth disorders) | 1
TINNITUS (Ear and labyrinth disorders) | 1
TYMPANIC MEMBRANE PERFORATION (Ear and labyrinth disorders) | 1
VERTIGO (Ear and labyrinth disorders) | 3
HYPERPARATHYROIDISM (Endocrine disorders) | 2
CONJUNCTIVAL HAEMORRHAGE (Eye disorders) | 1
CONJUNCTIVITIS (Eye disorders) | 1
EYE INFLAMMATION (Eye disorders) | 1
LACRIMATION INCREASED (Eye disorders) | 1
RETINOPATHY HYPERTENSIVE (Eye disorders) | 2
UVEITIS (Eye disorders) | 1
VISION BLURRED (Eye disorders) | 1
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 3
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 2
CONSTIPATION (Gastrointestinal disorders) | 3
DIARRHOEA (Gastrointestinal disorders) | 13
DRY MOUTH (Gastrointestinal disorders) | 1
DYSPEPSIA (Gastrointestinal disorders) | 1
DYSPHAGIA (Gastrointestinal disorders) | 1
ENTERITIS (Gastrointestinal disorders) | 2
GASTROINTESTINAL DISORDER (Gastrointestinal disorders) | 1
GASTROINTESTINAL PAIN (Gastrointestinal disorders) | 1
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 1
GINGIVAL HYPERTROPHY (Gastrointestinal disorders) | 1
MOUTH ULCERATION (Gastrointestinal disorders) | 1
NAUSEA (Gastrointestinal disorders) | 5
ODYNOPHAGIA (Gastrointestinal disorders) | 2
STOMATITIS (Gastrointestinal disorders) | 1
VOMITING (Gastrointestinal disorders) | 6
ASTHENIA (General disorders) | 6
CALCINOSIS (General disorders) | 1
CATHETER SITE DISCHARGE (General disorders) | 1
CATHETER SITE ERYTHEMA (General disorders) | 1
CATHETER SITE PRURITUS (General disorders) | 1
CHEST DISCOMFORT (General disorders) | 1
CHEST PAIN (General disorders) | 2
CHILLS (General disorders) | 1
DEVICE OCCLUSION (General disorders) | 1
FATIGUE (General disorders) | 3
IMPAIRED HEALING (General disorders) | 1
INFLUENZA LIKE ILLNESS (General disorders) | 1
MALAISE (General disorders) | 1
MEDICAL DEVICE COMPLICATION (General disorders) | 2
OEDEMA (General disorders) | 2
OEDEMA PERIPHERAL (General disorders) | 9
PYREXIA (General disorders) | 7
CHOLECYSTITIS (Hepatobiliary disorders) | 1
CHOLELITHIASIS (Hepatobiliary disorders) | 1
CHOLESTASIS (Hepatobiliary disorders) | 2
HEPATOCELLULAR INJURY (Hepatobiliary disorders) | 1
ASYMPTOMATIC BACTERIURIA (Infections and infestations) | 1
BACTERIAL INFECTION (Infections and infestations) | 1
BACTERIURIA (Infections and infestations) | 1
BK VIRUS INFECTION (Infections and infestations) | 1
BRONCHITIS (Infections and infestations) | 5
BRONCHITIS VIRAL (Infections and infestations) | 1
CATHETER SITE INFECTION (Infections and infestations) | 1
CYSTITIS (Infections and infestations) | 1
DENTAL GANGRENE (Infections and infestations) | 1
DEVICE RELATED INFECTION (Infections and infestations) | 1
DEVICE RELATED SEPSIS (Infections and infestations) | 1
EAR INFECTION (Infections and infestations) | 1
ERYSIPELAS (Infections and infestations) | 1
FOLLICULITIS (Infections and infestations) | 1
GASTROENTERITIS (Infections and infestations) | 3
GENITAL INFECTION FUNGAL (Infections and infestations) | 1
HERPES ZOSTER (Infections and infestations) | 1
INFECTION (Infections and infestations) | 1
INFLUENZA (Infections and infestations) | 2
LARYNGITIS (Infections and infestations) | 1
LUNG INFECTION (Infections and infestations) | 1
LYMPHANGITIS (Infections and infestations) | 1
NASOPHARYNGITIS (Infections and infestations) | 8
ONYCHOMYCOSIS (Infections and infestations) | 1
ORAL FUNGAL INFECTION (Infections and infestations) | 1
ORAL HERPES (Infections and infestations) | 3
OTITIS MEDIA (Infections and infestations) | 1
PHARYNGITIS (Infections and infestations) | 1
PULMONARY SEPSIS (Infections and infestations) | 1
PYELONEPHRITIS (Infections and infestations) | 1
RESPIRATORY TRACT INFECTION (Infections and infestations) | 1
RHINITIS (Infections and infestations) | 3
SINUSITIS (Infections and infestations) | 2
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 2
TINEA PEDIS (Infections and infestations) | 1
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1
URINARY TRACT INFECTION (Infections and infestations) | 7
VAGINITIS BACTERIAL (Infections and infestations) | 1
VIRAL INFECTION (Infections and infestations) | 2
ARTERIOVENOUS FISTULA SITE COMPLICATION (Injury, poisoning and procedural complications) | 1
CONTUSION (Injury, poisoning and procedural complications) | 1
FOOT FRACTURE (Injury, poisoning and procedural complications) | 1
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 1
PROCEDURAL COMPLICATION (Injury, poisoning and procedural complications) | 1
SHUNT MALFUNCTION (Injury, poisoning and procedural complications) | 1
SKELETAL INJURY (Injury, poisoning and procedural complications) | 1
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 1
WOUND (Injury, poisoning and procedural complications) | 1
BLOOD PRESSURE INCREASED (Investigations) | 1
CARDIAC MURMUR (Investigations) | 2
EOSINOPHIL COUNT INCREASED (Investigations) | 2
FREE HAEMOGLOBIN PRESENT (Investigations) | 1
LIVER FUNCTION TEST ABNORMAL (Investigations) | 1
PLATELET COUNT DECREASED (Investigations) | 2
URINE PROTEIN/CREATININE RATIO INCREASED (Investigations) | 1
WEIGHT DECREASED (Investigations) | 1
WHITE BLOOD CELL COUNT INCREASED (Investigations) | 1
ACIDOSIS (Metabolism and nutrition disorders) | 2
DECREASED APPETITE (Metabolism and nutrition disorders) | 1
DEHYDRATION (Metabolism and nutrition disorders) | 1
ELECTROLYTE IMBALANCE (Metabolism and nutrition disorders) | 1
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 1
HYPERCREATININAEMIA (Metabolism and nutrition disorders) | 2
HYPERKALAEMIA (Metabolism and nutrition disorders) | 4
HYPERPHOSPHATAEMIA (Metabolism and nutrition disorders) | 5
HYPERURICAEMIA (Metabolism and nutrition disorders) | 1
HYPERVOLAEMIA (Metabolism and nutrition disorders) | 2
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 3
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 1
HYPOKALAEMIA (Metabolism and nutrition disorders) | 4
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 1
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 4
IRON DEFICIENCY (Metabolism and nutrition disorders) | 1
METABOLIC ACIDOSIS (Metabolism and nutrition disorders) | 1
OVERWEIGHT (Metabolism and nutrition disorders) | 1
TYPE 2 DIABETES MELLITUS (Metabolism and nutrition disorders) | 1
VITAMIN D DEFICIENCY (Metabolism and nutrition disorders) | 4
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 8
BACK PAIN (Musculoskeletal and connective tissue disorders) | 3
BONE PAIN (Musculoskeletal and connective tissue disorders) | 1
CHONDROCALCINOSIS (Musculoskeletal and connective tissue disorders) | 1
HAEMARTHROSIS (Musculoskeletal and connective tissue disorders) | 1
JOINT EFFUSION (Musculoskeletal and connective tissue disorders) | 1
JOINT STIFFNESS (Musculoskeletal and connective tissue disorders) | 1
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 1
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 2
MYALGIA (Musculoskeletal and connective tissue disorders) | 4
NECK PAIN (Musculoskeletal and connective tissue disorders) | 2
OSTEOPENIA (Musculoskeletal and connective tissue disorders) | 1
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 2
RHABDOMYOLYSIS (Musculoskeletal and connective tissue disorders) | 1
PARATHYROID TUMOUR BENIGN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
AMNESIA (Nervous system disorders) | 1
DIZZINESS (Nervous system disorders) | 2
HEADACHE (Nervous system disorders) | 15
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 1
MIGRAINE (Nervous system disorders) | 2
PARAESTHESIA (Nervous system disorders) | 3
POLYNEUROPATHY (Nervous system disorders) | 1
PRESYNCOPE (Nervous system disorders) | 1
SCIATICA (Nervous system disorders) | 1
SYNCOPE (Nervous system disorders) | 1
TREMOR (Nervous system disorders) | 1
AGITATION (Psychiatric disorders) | 1
ANXIETY (Psychiatric disorders) | 4
DEPRESSED MOOD (Psychiatric disorders) | 2
DEPRESSION (Psychiatric disorders) | 3
INSOMNIA (Psychiatric disorders) | 5
NIGHTMARE (Psychiatric disorders) | 1
ANURIA (Renal and urinary disorders) | 1
DYSURIA (Renal and urinary disorders) | 1
HAEMATURIA (Renal and urinary disorders) | 1
PROTEINURIA (Renal and urinary disorders) | 5
RENAL FAILURE ACUTE (Renal and urinary disorders) | 1
RENAL FAILURE CHRONIC (Renal and urinary disorders) | 2
RENAL IMPAIRMENT (Renal and urinary disorders) | 6
RENAL VESSEL DISORDER (Renal and urinary disorders) | 1
TUBULOINTERSTITIAL NEPHRITIS (Renal and urinary disorders) | 1
URINE ABNORMALITY (Renal and urinary disorders) | 1
VESICOURETERIC REFLUX (Renal and urinary disorders) | 1
AMENORRHOEA (Reproductive system and breast disorders) | 2
ATROPHIC VULVOVAGINITIS (Reproductive system and breast disorders) | 1
BREAST CYST (Reproductive system and breast disorders) | 1
DYSMENORRHOEA (Reproductive system and breast disorders) | 2
ENDOMETRIOSIS (Reproductive system and breast disorders) | 1
HAEMATOSPERMIA (Reproductive system and breast disorders) | 1
METRORRHAGIA (Reproductive system and breast disorders) | 1
COUGH (Respiratory, thoracic and mediastinal disorders) | 7
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 5
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 2
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1
NASAL SEPTUM DEVIATION (Respiratory, thoracic and mediastinal disorders) | 1
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 3
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 2
PULMONARY CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1
RHINITIS ALLERGIC (Respiratory, thoracic and mediastinal disorders) | 1
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 2
SNORING (Respiratory, thoracic and mediastinal disorders) | 1
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 1
ALOPECIA (Skin and subcutaneous tissue disorders) | 5
DERMATITIS (Skin and subcutaneous tissue disorders) | 1
ECZEMA (Skin and subcutaneous tissue disorders) | 2
ERYTHEMA (Skin and subcutaneous tissue disorders) | 2
INTERTRIGO (Skin and subcutaneous tissue disorders) | 1
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 1
PETECHIAE (Skin and subcutaneous tissue disorders) | 1
PHOTOSENSITIVITY REACTION (Skin and subcutaneous tissue disorders) | 1
PRURITUS (Skin and subcutaneous tissue disorders) | 4
PURPURA (Skin and subcutaneous tissue disorders) | 2
RASH (Skin and subcutaneous tissue disorders) | 4
RASH ERYTHEMATOUS (Skin and subcutaneous tissue disorders) | 1
RASH PRURITIC (Skin and subcutaneous tissue disorders) | 2
SKIN DISCOLOURATION (Skin and subcutaneous tissue disorders) | 1
URTICARIA (Skin and subcutaneous tissue disorders) | 2
DEEP VEIN THROMBOSIS (Vascular disorders) | 1
HAEMATOMA (Vascular disorders) | 3
HOT FLUSH (Vascular disorders) | 1
HYPERTENSION (Vascular disorders) | 5
HYPOTENSION (Vascular disorders) | 7
STEAL SYNDROME (Vascular disorders) | 1
THROMBOPHLEBITIS (Vascular disorders) | 1
VENOUS THROMBOSIS (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Participation in this multicenter study involved a commitment to publish the data from the study in a cooperative publication prior to release of study results on an individual basis.